CLINICAL TRIAL: NCT06657755
Title: A Study to Evaluate ENPP1 Expression and Its Role in Immune Evasion and Chemoresistance in Bladder Cancer
Brief Title: Evaluation of ENPP1 Expression and Immune Response in Bladder Cancer Patients
Acronym: ENPP1-BC
Status: Completed | Type: Observational
Sponsor: Lanzhou University Second Hospital (Other)
Responsible Party: Principal Investigator, Chengyu You, Lanzhou University Second Hospital, Lanzhou University Second Hospital
Other Study IDs: 2024A-948; D2024-686 (Other: Lanzhou University Second Hospital)
Record Dates: First submitted 2024-10-21; First posted 2024-10-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Bladder (Urothelial, Transitional Cell) Cancer
Keywords: ENPP1; bladder cancer; biomarker; prognosis; immune infiltration
MeSH Terms: conditions — Neoplasms; Urinary Bladder Neoplasms | interventions — Immunohistochemistry

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Tissue samples, blood samples, and other relevant biological specimens will be retained for future analysis, including potential DNA extraction for genetic studies.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Immunohistochemistry — This intervention will specifically focus on evaluating the role of ENPP1 in bladder cancer patients, distinguishing it from other interventions by targeting immune evasion and chemoresistance pathways. The intervention will include a combination of targeted molecular therapies and immunotherapy, aimed at assessing the therapeutic potential of ENPP1 inhibition in improving treatment outcomes for bladder cancer patients. This differs from previous studies by integrating advanced biomarker analysis and personalized treatment approaches based on ENPP1 expression levels.

SUMMARY:
This study aims to investigate the role of ENPP1 in bladder cancer (BC), specifically focusing on its impact on immune evasion, chemoresistance, and prognosis. The study will analyze gene expression data from clinical samples and use various laboratory techniques, including RNA sequencing, qRT-PCR, and immunohistochemistry, to assess ENPP1's expression levels. In addition, the research will explore the relationship between ENPP1 and immune cell infiltration, along with its correlation with patient survival outcomes. By identifying ENPP1's contribution to cancer progression and treatment resistance, the study aims to discover potential therapeutic targets for improving bladder cancer treatment strategies.

DETAILED DESCRIPTION:
This study is designed to comprehensively explore the role of ENPP1 (Ectonucleotide Pyrophosphatase/Phosphodiesterase 1) in bladder cancer (BC) development and progression. ENPP1 has been implicated in various cancers, with evidence suggesting its involvement in immune evasion, chemoresistance, and poor prognosis. However, its specific function in bladder cancer remains unclear. This research will analyze clinical samples, including tumor tissues and normal adjacent tissues, to evaluate ENPP1 expression through a combination of advanced laboratory techniques such as RNA sequencing, quantitative real-time PCR (qRT-PCR), Western blotting, immunohistochemistry (IHC), and immunofluorescence.

Furthermore, the study will investigate the association between ENPP1 expression and key clinical parameters, including tumor stage, grade, lymph node involvement, metastasis, and patient survival outcomes. Through bioinformatics tools, immune infiltration analysis will be conducted to assess the impact of ENPP1 on immune cells such as CD8+ T cells, dendritic cells, and M2 macrophages, which are crucial in the tumor microenvironment.

The research will also explore the correlation between ENPP1 expression and resistance to common chemotherapeutic agents, particularly gemcitabine and cytarabine, using drug sensitivity data from public databases. By identifying the molecular mechanisms by which ENPP1 influences immune responses and chemoresistance, the study aims to provide valuable insights into potential therapeutic targets for bladder cancer treatment. Ultimately, this research may contribute to the development of personalized therapies for bladder cancer patients based on ENPP1 expression.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older.
* Histologically confirmed diagnosis of bladder cancer.
* Measurable disease as per RECIST criteria.
* Adequate organ function as defined by laboratory tests (e.g., liver, kidney, and hematologic function).
* ENPP1 expression level determined via biopsy or previous analysis.
* Written informed consent provided.

Exclusion Criteria:

* History of other malignancies within the past 5 years, excluding non-melanoma skin cancer or in situ carcinoma.
* Prior treatment with ENPP1 inhibitors or similar targeted therapies.
* Active or uncontrolled infections.
* Pregnant or breastfeeding women.
* Known autoimmune disorders or conditions requiring immunosuppressive therapy.
* Inability to comply with the study protocol or procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adult patients aged 18 years or older with a confirmed diagnosis of bladder cancer. Participants will be recruited from oncology clinics and hospitals, and all eligible individuals must have measurable disease as defined by RECIST criteria. Both male and female participants will be included, with no restrictions based on ethnicity or socioeconomic background. Participants will be required to provide informed consent and meet the inclusion criteria related to health status and prior treatments.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-20 (Actual)

PRIMARY OUTCOMES:
ENPP1 Expression Levels in Bladder Cancer Patients | 2024.1-2024.6
  The primary outcome will measure the expression levels of ENPP1 in bladder cancer tissues compared to adjacent normal tissues, and its correlation with clinical outcomes such as overall survival (OS) and progression-free survival (PFS).

CONTACTS AND LOCATIONS:
Overall Officials: Zhilong Dong, MD, Study Director — Lanzhou University Second Hospital
Locations (1):
- Lanzhou University Second Hospital, Lanzhou, Gansu, China

IPD SHARING:
Plan to Share IPD: No
We do not plan to share individual participant data (IPD) with other researchers due to the sensitive nature of the clinical data involved. However, aggregated data and relevant findings from the study will be published in peer-reviewed journals to contribute to the scientific community.

REFERENCES:
- [Background] An Y, Zhu J, Xie Q, Feng J, Gong Y, Fan Q, Cao J, Huang Z, Shi W, Lin Q, Wu L, Yang C, Ji T. Tumor Exosomal ENPP1 Hydrolyzes cGAMP to Inhibit cGAS-STING Signaling. Adv Sci (Weinh). 2024 May;11(20):e2308131. doi: 10.1002/advs.202308131. Epub 2024 Mar 18. PMID 38498770
- [Background] Li J, Duran MA, Dhanota N, Chatila WK, Bettigole SE, Kwon J, Sriram RK, Humphries MP, Salto-Tellez M, James JA, Hanna MG, Melms JC, Vallabhaneni S, Litchfield K, Usaite I, Biswas D, Bareja R, Li HW, Martin ML, Dorsaint P, Cavallo JA, Li P, Pauli C, Gottesdiener L, DiPardo BJ, Hollmann TJ, Merghoub T, Wen HY, Reis-Filho JS, Riaz N, Su SM, Kalbasi A, Vasan N, Powell SN, Wolchok JD, Elemento O, Swanton C, Shoushtari AN, Parkes EE, Izar B, Bakhoum SF. Metastasis and Immune Evasion from Extracellular cGAMP Hydrolysis. Cancer Discov. 2021 May;11(5):1212-1227. doi: 10.1158/2159-8290.CD-20-0387. Epub 2020 Dec 28. PMID 33372007
- [Background] Bageritz J, Puccio L, Piro RM, Hovestadt V, Phillips E, Pankert T, Lohr J, Herold-Mende C, Lichter P, Goidts V. Stem cell characteristics in glioblastoma are maintained by the ecto-nucleotidase E-NPP1. Cell Death Differ. 2014 Jun;21(6):929-40. doi: 10.1038/cdd.2014.12. Epub 2014 Feb 14. PMID 24531536
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- See also: Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries — https://pubmed.ncbi.nlm.nih.gov/33538338/
- See also: Stem cell characteristics in glioblastoma are maintained by the ecto-nucleotidase E-NPP1 — https://pmc.ncbi.nlm.nih.gov/articles/PMC4013511/
- See also: Metastasis and Immune Evasion from Extracellular cGAMP Hydrolysis — https://pmc.ncbi.nlm.nih.gov/articles/PMC8102348/
- See also: Tumor Exosomal ENPP1 Hydrolyzes cGAMP to Inhibit cGAS-STING Signaling — https://pmc.ncbi.nlm.nih.gov/articles/PMC11132070/